CLINICAL TRIAL: NCT07380542
Title: Dynamic Magnesium Replacement Strategies and 28-Day All-Cause Mortality in Non-Cardiac Critically Ill Patients With Hypomagnesemia: A Target Trial Emulation Using the MIMIC-IV Database (2008-2019)
Brief Title: Dynamic Magnesium Replacement Strategies and 28-Day Mortality in Non-Cardiac Critically Ill Patients With Hypomagnesemia: A Target Trial Emulation
Status: Completed | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Han Chen, Professor, Fujian Provincial Hospital
Other Study IDs: HChen-MgReple2025
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hypomagnesemia
Keywords: Magnesium Replacement Therapy; 28-Day Mortality; Intensive Care Unit Patients; Target Trial Emulation; Retrospective Cohort Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Never Treat Group: Patients with hypomagnesemia who received no magnesium replacement therapy during their ICU stay, regardless of daily serum magnesium levels
- Always Treat Group: Patients with hypomagnesemia who received daily magnesium replacement therapy during their ICU stay, regardless of daily serum magnesium levels
- Dynamic Treat Group: Patients with hypomagnesemia who received magnesium replacement therapy only on days when their daily serum magnesium level was <1.7 mg/dL during their ICU stay

SUMMARY:
This study looks at how different ways of giving magnesium (a nutrient) affect the risk of death within 28 days for adults with low magnesium levels who are in the intensive care unit (ICU) for non-heart-related reasons. We will use data from past ICU patients (2008-2019) to compare three approaches:

No magnesium treatment (even if levels are low); Daily magnesium treatment (regardless of daily levels); Dynamic treatment (only giving magnesium when daily tests show low levels). The goal is to find out which strategy is safest and most effective for this group of patients.

DETAILED DESCRIPTION:
This is a target trial emulation (a type of observational study that mimics a clinical trial) using data from the Medical Information Mart for Intensive Care IV (MIMIC-IV) database (2008-2019).

Inclusion criteria: Adults (≥18 years) admitted to the ICU, with serum magnesium <1.7 mg/dL within 72 hours of admission, and no history of heart disease or cardiac surgery.

Sample size: 12,887 patients. Interventions (simulated): Three magnesium replacement strategies (Never Treat, Always Treat, Dynamic Treat).

Outcome: 28-day all-cause mortality (death from any cause). Analysis methods: We will use the G-formula (to handle time-varying factors that could affect results) and sensitivity analyses to check if findings are reliable.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Admitted to the Intensive Care Unit (ICU).
3. Developed hypomagnesemia (Serum Magnesium < 1.7 mg/dL) within the first 72 hours of ICU admission.

Exclusion Criteria:

1. Admitted due to cardiac or cardiosurgical causes (e.g., Cardiac Surgery Recovery Unit, CCU, CVICU).
2. Underwent cardiac surgery during hospitalization (identified by ICD-9/10 procedure codes).
3. Primary discharge diagnosis of major cardiac conditions (e.g., myocardial infarction, heart failure, arrhythmias).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult (≥18 years) non-cardiac critically ill patients with hypomagnesemia (serum magnesium < 1.7 mg/dL) within 72 hours of ICU admission, identified from the MIMIC-IV (version 3.1) database (2008-2019). Patients with cardiac-related admission or missing key data are excluded. The population represents a diverse cohort of non-cardiac ICU patients (e.g., respiratory, gastrointestinal, neurological etiologies) to evaluate the association between dynamic magnesium replacement strategies and 28-day mortality.
Sampling Method: Non-Probability Sample
Enrollment: 12887 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
28-Day All-Cause Mortality | 28 days after t0
  Death from any cause within 28 days after t0 (t0 = the first time serum magnesium <1.7 mg/dL is detected within 72 hours of hospital admission)

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) cannot be shared because the study uses data from the MIMIC-IV database, which requires researchers to complete mandatory training and obtain independent authorization from the MIMIC-IV Data Access Committee. IPD is not owned by the study team; qualified researchers may access the data directly via the official MIMIC-IV application process (https://mimic.mit.edu/).

REFERENCES:
- [Background] Hernan MA, Robins JM. Using Big Data to Emulate a Target Trial When a Randomized Trial Is Not Available. Am J Epidemiol. 2016 Apr 15;183(8):758-64. doi: 10.1093/aje/kwv254. Epub 2016 Mar 18. PMID 26994063
- [Background] Johnson AEW, Bulgarelli L, Shen L, Gayles A, Shammout A, Horng S, Pollard TJ, Hao S, Moody B, Gow B, Lehman LH, Celi LA, Mark RG. MIMIC-IV, a freely accessible electronic health record dataset. Sci Data. 2023 Jan 3;10(1):1. doi: 10.1038/s41597-022-01899-x. PMID 36596836

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT07380542/Prot_SAP_000.pdf